CLINICAL TRIAL: NCT06484257
Title: Comparison Between Myopia Versus Hypermetropia With Progressive Addition Lenses in Computer Users
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/732
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Myopia; Hypermetropia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myopia (Active Comparator)
  Interventions: Behavioral: Myopia
- Hypermetropia (Other)
  Interventions: Other: Hypermetropia

INTERVENTIONS:
Behavioral: Myopia — Participants in this arm would receive progressive addition lenses specifically designed to correct myopia. These lenses would typically have a prescription for correcting nearsightedness (myopia) in addition to any other vision corrections needed, such as astigmatism correction and presbyopia. The participants would wear these lenses while using computers according to the study protocol.
  Arms: Myopia
Other: Hypermetropia — Participants in this arm would receive progressive addition lenses specifically designed to correct hypermetropia. These lenses would typically have a prescription for correcting farsightedness (hypermetropia) in addition to any other vision corrections needed, such as astigmatism correction and presbyopia. The participants would wear these lenses while using computers according to the study protocol.
  Arms: Hypermetropia

SUMMARY:
This study examines how myopia (nearsightedness) and hyperopia (farsightedness) affect the use of progressive addition lenses (PALs) for computer users. PALs offer a range of vision correction within one lens, ideal for presbyopia (age-related near focusing difficulty). We'll compare visual comfort, eye strain, and user preference for PALs between myopic and hyperopic individuals while focusing on computer screens.

DETAILED DESCRIPTION:
The research will also consider if general-purpose PALs differ from computer-specific PALs in these user groups, and how presbyopia progression might influence PAL effectiveness for each condition. This information can help eye doctors recommend the most suitable PAL design for computer users with myopia or hyperopia.

ELIGIBILITY:
Inclusion Criteria:

* The age of Participant will be 40 to 55 years
* Participant diagnosed with myopia having -0.50 to -3.00DS and astigmatism up to -0.75DC
* Patient diagnosed with Hypermetropia having +050 to +3.00 DS and Astigmatism up to +0.75DC
* Presbyopia addition will range from +1.00 to +2.50 DS
* Participants who have worked more than 4 hours on the computer screen.
* Participants who will be already progressive users and first-time users.
* Patients with no Ocular disease.

Exclusion Criteria:

* Participants with Pre Presbyopia and above 55 years of age
* Participants with significant ocular disease.
* Participants with uncontrolled diabetes and hypertension
* Participants who will not be willing for PAL,s
* Participants with more than 0.75 astigmatism
* Participants with known allergies and sensitivity.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 12 Months
  Assessing visual acuity at different distances, including distance vision (for activities such as viewing the computer screen) and near vision (for reading text on the screen), while wearing progressive addition lenses.
Subjective Visual Comfort | 12 months
  Using standardized questionnaires or subjective ratings from participants to assess their comfort level while using computers with progressive addition lenses.
Visual Fatigue | 12 months
  Assessing the level of visual fatigue experienced by participants during or after prolonged computer use with the progressive addition lenses. This could involve subjective ratings of eye strain, tiredness, or discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- The Keratoconus center, Eye 2 Eye Optometrists, 13 D valencia housing society, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No